CLINICAL TRIAL: NCT03035500
Title: Long-term Follow-up After Prostate Cancer
Brief Title: Long-Term Follow-Up in Patients With Prostate Cancer After Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 07101; NCI-2017-00090 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 07101 (Other: City of Hope Medical Center)
Record Dates: First submitted 2017-01-25; First posted 2017-01-30 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cancer Survivor; Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive Care (long-term follow-up) (Experimental): Patients undergo long-term follow-up and receive a written survivorship care plan including comprehensive health evaluation and health education beginning 1 year post surgery.
  Interventions: Other: Educational Intervention; Other: Laboratory Biomarker Analysis; Other: Long-term Follow-up; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive health education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Long-term Follow-up — Undergo long-term follow-up using survivorship care plan
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well a long-term follow-up works in patients with prostate cancer after surgery. Long-term follow-up data may serve as a resource to help ask clinical questions, describe health-related quality of life and long-term complications related, and facilitate future studies focusing on interventions to improve health status and health-related quality of life in prostate cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide comprehensive long-term follow-up care to prostate cancer survivors at the City of Hope who underwent definitive surgical therapy.

II. To use the information obtained from follow-up of prostate cancer survivors who underwent definitive surgical therapy to serve as a resource that will help answer clinical questions, generate and test hypotheses, describe the incidence of long-term complications, and facilitate future studies focusing on interventions for long-term complications of prostate cancer and its therapy.

III. To use the information gained from follow-up of prostate cancer survivors who underwent definitive surgical therapy to describe health-related quality of life (HRQL) concerns and to serve as a resource to facilitate future studies focusing on interventions to improve health status and HRQL in prostate cancer survivors.

OUTLINE:

Patients undergo long-term follow-up and receive a written survivorship care plan including comprehensive health evaluation and health education beginning 1 year post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer
* Treated with a definitive surgical procedure at City of Hope
* At least one year post surgical treatment for prostate cancer
* No history of recurrent, progressive, or metastatic disease
* Currently stable disease or no evidence of disease
* No prior treatment of prostate cancer with radiation or chemotherapy
* No history of other urologic cancer (e.g., bladder cancer, renal cell carcinoma) in addition to prostate cancer

  * Note: Patients who develop recurrence while participating in the Prostate Cancer Survivorship Clinic will be referred back to their urologist and may resume participation in the Survivorship Clinic when deemed appropriate by their treating physician

Exclusion Criteria:

* Current treatment with testosterone replacement or androgen deprivation therapy
* Treatment for another noncutaneous cancer within the past 2 years

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2008-07-23 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
HRQL assessed using Expanded Prostate Cancer Index Composite | Up to 10 years
  Linear mixed effects models can be used to estimate long-term trends and examine the effects of baseline and concomitant factors on these trends.
HRQL assessed using Sexual Health Inventory for Men | Up to 10 years
  Linear mixed effects models can be used to estimate long-term trends and examine the effects of baseline and concomitant factors on these trends.
Incidence rates of the study end-points | Up to 10 years
  Incidence rates of the study end-points that may be associated with original diagnosis or treatment received, and delineation of temporal changes in serial measurements and their relationship to time-invariant characteristics such as original diagnosis, race, and education and time-varying characteristics such as age and body mass index will be estimated. Incidence rates may be compared with national standards adjusted for key demographic variables and between patient subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Saro Armenian, DO, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States